CLINICAL TRIAL: NCT05233657
Title: An Evaluation of Safety, Tolerability and Pharmacokinetics of Single Oral Dose of JX11502MA Capsule on Healthy Human: A Phase Ia, Single Center, Randomized Clinical Trial
Brief Title: A Safety，Tolerability and Pharmacokinetics Clinical Trial of JX11502MA Capsule
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Jingxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JX11502MA-I-01
Record Dates: First submitted 2021-12-12; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2021-12

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- JX11502MA 0.25mg、0.5mg、1mg、2mg、3mg、6mg、8mg (Experimental): Participants received JX11502MA capsule 0.25mg、0.5mg、1mg、2mg、3mg、6mg、8mg orally administration once, once on an empty stomach in the morning, with about 240ml of warm water.
  Interventions: Drug: JX11502MA
- Placebo 0.25mg、0.5mg、1mg、2mg、3mg、6mg、8mg (Placebo Comparator): Participants received placebo capsule 0.25mg、0.5mg、1mg、2mg、3mg、6mg、8mg orally administration once, once on an empty stomach in the morning, with about 240ml of warm water..
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JX11502MA — Oral capsule
  Arms: JX11502MA 0.25mg、0.5mg、1mg、2mg、3mg、6mg、8mg
Drug: Placebo — Oral capsule
  Arms: Placebo 0.25mg、0.5mg、1mg、2mg、3mg、6mg、8mg

SUMMARY:
The purpose of this study is to investigate the safety, tolerability and pharmacokinetic characteristics of JX11502MA capsule on healthy human, and to explore the relationship between the dose, pharmacokinetic parameters and safety of JX11502MA capsule，so as to provide basis for the follow-up clinical trials (multi-dose tolerability, pharmacokinetics and phase II trial, etc.).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects;
2. The age is between 18 and 45 years old (including the margin value);
3. Male ≥50 kg, female ≥45 kg, the body mass index (BMI) of subjects ranged from 19 to 28 kg/m2 (including the boundary value);
4. Be able to understand informed consent, voluntarily participate in clinical trials and sign informed consent;
5. Be able to complete the experiment according to the research plan. Those who do not meet one of the above conditions shall not be selected as subjects.

Exclusion Criteria:

1. The researcher judged that the subjects has current and past medical diseases or dysfunction history that may affect clinical trial, including but not limited to diseases of central nervous system, cardiovascular system, respiratory system, digestive system, urinary system, endocrine system and blood system;
2. Suffering from mental illness or previous history of mental illness;
3. Have a history of ophthalmic diseases, such as abnormal color vision, retinitis pigmentosa, macular degeneration, etc;
4. Have a history of malignant tumors or other diseases that are not suitable for clinical trials;
5. Any surgical situation or condition that may significantly affect the absorption, distribution, metabolism and excretion of drugs, or any surgical condition that may harm the subjects participating in this trial; Such as gastrointestinal surgery history (gastrectomy, gastrointestinal anastomosis, intestinal resection, etc.), urinary tract obstruction or dysuria, gastroenteritis, gastrointestinal ulcer, gastrointestinal bleeding history, etc.;
6. Those who have allergic history of similar drug, allergic disease history or allergic constitution history;
7. Those who are addicted to tobacco within one year before screening and smoke more than 10 cigarettes or the same amount of tobacco average every day;
8. Those who are addicted to alcohol within one year before screening, and the average weekly alcohol intake exceeds 14 units (1 unit =285 mL beer or 25 mL spirits or 150 mL wine) or those who are positive for alcohol breath test;
9. Those who have a history of drug and drug abuse within one year before screening, or those who are positive for urine drug screening;
10. Physical examination, present medical history and vital signs, which are judged by researchers to be abnormal and have a clinical significance;
11. Resting pulse rate < 55 beats/min or > 100 beats/min; Systolic pressure < 90 mmHg or > 140 mmHg, diastolic pressure < 60 mmHg or > 90 mmHg;
12. Abnormal and has a clinical significance of 12-lead electrocardiogram (ECG) examination result judged by researchers; Or appears following ECG abnormalities: PR interval > 220 ms, QRS complex web time limit > 120 ms, long QT syndrome (QTC > 450 ms);
13. Family history of sudden cardiac death (Lower than 40 years old);
14. Abnormal and have clinical significance of blood routine examination and urine routine examination;
15. Exceeded the normal limit of aspartate transferase (AST), alanine transferase (ALT), creatinine (Cr) and urea nitrogen (BUN) .
16. Subjects with positive hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), HIV antibody (HIV-Ab) and syphilis seroreaction (TRUST);
17. Pregnant and lactating women, or those who have the ability to conceive/pregnant, don't agree to adopt recognize effective methods of contraception during the study period and within 3 months after stopping treatment;
18. Those who take any drugs within 2 weeks before before enrolling the trial, including prescription drugs and over-the-counter drugs;
19. Blood donation or blood loss ≥200 mL within 3 months before enrolling, or history of using blood products;
20. Participated any clinical trial within 3 months before enrolling the trial;
21. Those who have a history of surgery within 3 months before enrollment, or haven't recover from surgery, or have expected surgical plan during the trial;
22. Don't agree to comply with the following conditions during the trial: prohibit the use of alcohol, tobacco or caffeinated beverages and avoid strenuous exercise;
23. Person those are directly related to this trial;
24. Researcher decide, subjects those are non-suitable to participate in this trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2020-01-04 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
The incidence rate of adverse reactions | Day（1）-Day（7）
  Count the number of subjects with adverse reactions during the trial and calculate the incidence of adverse reactions（Number of subjects with adverse reactions / total number of subjects* 100%）.The adverse reactions include drowsiness、weakness hiccup、vomit、anorexia、nausea、insomnia、dry mouth、dizzy and stomach distention

SECONDARY OUTCOMES:
Cmax | Day（1）-Day（7）
  Maximum Serum Concentration of the parent drug
Tmax | Day（1）-Day（7）
  Time to Reach the Maximum Serum Concentration of the parent drug
AUC | Day（1）-Day（7）
  Area Under the Serum Concentration-Time Curve of the parent drug
t1/2 | Day（1）-Day（7）
  Elimination half-life period

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu Y, He J, Huang Z, Li Y, Wu Y, Shen Y, Zhou Y, Bao C, Jin Z, Li H. Safety, tolerability, and pharmacokinetics of JX11502MA in Chinese healthy subjects: a first-in-human, randomized, double-blind, placebo-controlled study following single-dose administration. Expert Opin Investig Drugs. 2024 Jan;33(1):51-61. doi: 10.1080/13543784.2023.2291470. Epub 2024 Feb 12. PMID 38054696